CLINICAL TRIAL: NCT06980155
Title: Clinical Study of XP-005 Personalized Vaccine Alone or in Combination With Toripalimab to Prevent the Relapse of Acute Myeloid Leukemia After Consolidation Therapy
Brief Title: XP-005 Personalized Vaccine Alone or in Combination With Toripalimab for the Prevention of Relapse After Remission in Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Xinpu BioTechnology Company Limited (Unknown)
Responsible Party: Principal Investigator, Junmin Li, Head of hematology, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PCV002-XP005
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Neoantigen; Vaccines; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoantigen tumor vaccine monotherapy arm (Experimental): Dose Escalation Phase vaccine: 0.4mg, 0.8mg, 1 mg Dose Expansion Phase vaccine: MTD or 1mg
  Interventions: Biological: Personalized neoantigen tumor vaccine
- Neoantigen tumor vaccine and Toripalimab combination arm (Experimental): Dose Escalation Phase vaccine: 0.4mg, 0.8mg, 1 mg Dose Expansion Phase vaccine: MTD or 1 mg Toripalimab: 240mg/dose
  Interventions: Biological: Personalized neoantigen tumor vaccine; Biological: PD-1 inhibitor

INTERVENTIONS:
Biological: Personalized neoantigen tumor vaccine — Neoantigen tumor vaccine
Biological: PD-1 inhibitor — Toripalimab
  Arms: Neoantigen tumor vaccine and Toripalimab combination arm

SUMMARY:
The main objective of this study is to observe and evaluate the safety and tolerability of the XP-005 personalized tumor mRNA vaccine, either alone or in combination with toripalimab, for the treatment of acute myeloid leukemia patients who are in remission with minimal residual disease (MRD) positive but cannot undergo allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily signs the written informed consent form and is able to comply with the scheduled visits and related procedures specified in the protocol
2. Subject must be ≥ 18 years old, with no gender restrictions
3. The expected survival period is ≥3 months
4. Conforming to the World Health Organization (WHO) 2022 classification criteria for Acute Myeloid Leukemia (AML).
5. Subject has completed induction and consolidation chemotherapy and has achieved complete remission (CR), complete remission with partial hematologic recovery (CRh), or complete remission with incomplete hematologic recovery (CRi) according to the 2022 European LeukemiaNet (ELN) criteria. The patient does not meet the criteria for or has contraindications to stem cell transplantation.

   CR is defined as: bone marrow blasts <5%, absence of circulating blasts or blasts with Aure rods; absence of extramedullary disease, absolute neutrophil count (ANC) ≥1.0 × 10^9/L, and platelet count ≥100 × 10^9/L.

   CRh is defined as: ANC ≥0.5 × 10^9/L, and platelet count ≥50 × 10^9/L, otherwise all other CR criteria met CRi is defined as: All CR criteria except for ANC <1.0 × 10^9/L or platelet count <100 × 10^9/L. If both CRh and CRi are considered, CRi only includes patients who do not meet the criteria for CRh.
6. MRD positivity (①when using MFC, MRD is considered positive if the proportion of immunophenotypically abnormal cells among CD45+ cells is ≥0.01%; ② when using qPCR, MRD is considered positive if the NPM1 <3log10 reduction in BM.
7. NPM1 mutation classification as Type A, D, G, H, B, and J
8. The peripheral blood HLA typing is HLA-A02:01
9. The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score is 0-2
10. Subject must be willing to provide existing valid diagnostic evidence prior to treatment or undergo bone marrow aspiration and biopsy, and must also be willing to undergo bone marrow aspiration and biopsy after receiving treatment

Exclusion Criteria:

1. Copy number variants (CNVs) or loss of heterozygosity (LOH) in HLA-related genes or chromosomal regions were detected by genetic sequencing
2. Received chemotherapy, hormonal therapy, traditional Chinese medicine with anti-tumor indications, or other anti-tumor treatments within 4 weeks before the first dose (for mitomycin and nitrosoureas, within 6 weeks after the last dose), or within 5 half-lives of immunotherapy or molecular targeted therapy
3. Received tumor vaccines, cellular therapy, or planned to receive other vaccines within 4 weeks before the first dose
4. Subject who has undergone major surgery other than diagnostic or biopsy procedures within 4 weeks before the first dose, or who are expected to undergo major surgery during the study period
5. Uncontrolled central nervous system (CNS) lymphoma
6. Patients with extramedullary disease, or those deemed unsuitable for enrollment by the investigator
7. Eligible for allogeneic bone marrow or allogeneic stem cell transplantation at the time of Screening
8. Subject has previously undergone allogeneic hematopoietic stem cell transplantation or organ transplantation, or who is planned to undergo organ transplantation during this study
9. Within 7 days before treatment, laboratory tests show:

   1. AST (SGOT) / ALT (SGPT) > 3 ULN
   2. Total bilirubin > 2 ULN
   3. eGFR < 45 mL/min
   4. SpO2 < 95% without supplemental oxygen
10. DIC (Disseminated Intravascular Coagulation)
11. Active malignancy
12. A history of interstitial lung disease (ILD), pulmonary interstitial fibrosis, or stage III or higher chronic obstructive pulmonary disease (COPD)
13. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second- or third-degree atrioventricular block; corrected QTc interval > 450 milliseconds for males and > 470 milliseconds for females,
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events within 6 months before the first dose,
    3. New York Heart Association (NYHA) functional class ≥ III heart failure or left ventricular ejection fraction (LVEF) < 50%
14. Other severe and/or uncontrollable diseases, as determined by the investigator, that possibly affect the subject to participate in this study, including but not limited to:

    1. A history of severe drug allergy, or known allergy to any component of the tumor vaccine or toripalimab injection formulation; or a history of severe allergic reactions to other monoclonal antibodies,
    2. A history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases,
    3. Evidence of severe or uncontrollable liver or kidney disease,
    4. Poorly controlled hypertension, diabetes, etc.,
    5. Patients with active ulcers or gastrointestinal bleeding,
    6. Presence of severe infections requiring intravenous antibiotics or hospitalization; or uncontrolled active infections within 4 weeks before the first dose,
    7. Active syphilis infection
15. Hepatitis B surface antigen (HBsAg) positive with peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) levels above the upper limit of normal; hepatitis C virus antibody (HCV Ab) positive with HCV RNA levels above the upper limit of normal
16. Pregnant or breastfeeding women
17. Subject who has taken part in other clinical trials within 4 weeks before the first dose (excluding those who failed screening) or whom the investigator deems unsuitable for participation in the clinical trial for other reasons
18. Received systemic immunosuppressive therapy (excluding topical glucocorticoids) within 1 month before enrollment (e.g., >10 mg/d prednisone or equivalent)
19. Men and women of childbearing potential should agree to use non-pharmacological contraceptive measures from the time of signing the informed consent form until 3 months after the last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) & Maximum tolerated dose (MTD) | Day1 to Day21
Biologically Effective Dose (BED) | Day1 to Day21
  If MTD is not reached, BED will be used.
Percentage of Participants With Adverse Events (AEs) | Up to 52 weeks
  Percentage of Participants with Adverse Events (AEs) by Severity According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
MRD negativity rate | Up to 52 weeks
Degree of MRD decrease | Up to 52 weeks
Duration of MRD response | Up to 52 weeks
Recurrence-Free Survival (RFS) | Up to 52 weeks
Overall survival (OS) | Up to 52 weeks
  Overall Survival of XP005 Personalized mRNA Tumor Vaccine
Analysis of the levels of tumor neoantigen-specific CD4+ and CD8+ T lymphocytes and their correlation with therapeutic efficacy | Up to 52 weeks
Changes in lymphocyte subset levels and their correlation with therapeutic efficacy | Up to 52 weeks
Serum cytokine test | Up to 52 weeks
  IL-2、IL-6、IL-10、TNF-α、IFN-γ、IL-4、IL-5、IL-8、IL-12P70、IL-17
Peripheral blood TCR sequences and abundance | Up to 52 weeks
Single-cell sequencing results | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No